CLINICAL TRIAL: NCT05686460
Title: Comparison of the Effect of Hegu Point Ice Massage and Music on Pain and Comfort Levels in Dysmenorrhea
Brief Title: Effect of Hegu Point Ice Massage and Music in Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Sevgi Çetin, Research Assistant Dr, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CBU-PAKİSCETİN-1
Record Dates: First submitted 2023-01-02; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Primary Dysmenorrhea
Keywords: comfort; ice massage; music; pain; dysmenorrhea
MeSH Terms: conditions — Pain; Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The researcher gave each students a number in random. Then, they were divided into three groups by random sampling method using the Excel program. The students who were randomly assigned to the 1st group with the Excel program were determined as intervention group 1 (ice massage), the 2nd group students were intervention group 2 (music medicine), the 3rd group students were group 3 control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ice massage (Experimental): The application applied 2 minutes of ice massage 7 times at 15-second intervals. The procedure was performed once on the first day and once on the second day of menstruation.
  Interventions: Behavioral: ice massage
- music medicine (Experimental): Depending on their preference, each participant wearing personalized headphones was played instrumental music in the pre-menstruation period for 30 minutes. The procedure was performed once on the first day and once on the second day of menstruation.
  Interventions: Behavioral: music medicine
- control (No Intervention): On the first and second days of menstruation, their pain levels of were assessed 4 times: when the pain started (pre-test), and then 30, 60 and 90 minutes after the pain started.

INTERVENTIONS:
Behavioral: ice massage — After the students who met the sample selection criteria applied Student Information Form. On the first day of the participating students' menstruation, prior to the application (when the pain started), the Visual Analogue Scale (VAS), General Comfort Questionnaire (GCQ) and Dysmenorrhea Follow-up Form were filled in at the pre-test. The Hegu point of the participating students was detected with the acupuncture point finder. Ice cubes whose dimensions were 2x2x2 cm were wrapped with gauze and placed in a plastic bag. Vaseline® jelly was spread on the application area. The application applied 2 minutes of ice massage 7 times at 15-second intervals. The participants' pain levels were assessed three times, as soon as the application was over, 30 and 60 minutes after the application (Post-test).
  On the second day of menstruation, the participants were asked to fill in the VAS, GCQ, and Effects of Dysmenorrhea Scale (EDS).
  Arms: ice massage
Behavioral: music medicine — After the students who met the sample selection criteria applied Student Information Form. On the first day of the participating students' menstruation, prior to the application (when the pain started), the Visual Analogue Scale (VAS), General Comfort Questionnaire (GCQ) and Dysmenorrhea Follow-up Form were filled in at the pre-test. Depending on their preference, each participant wearing personalized headphones was played instrumental music in the pre-menstruation period for 30 minutes. The volume of the music was adjusted based on the verbal feedback or facial expressions of the students. The participants' pain levels were assessed three times, as soon as the application was over, 30 and 60 minutes after the application (Post-test). On the second day of menstruation, the participants were asked to fill in the VAS, GCQ, and Effects of Dysmenorrhea Scale (EDS).
  Arms: music medicine

SUMMARY:
Dysmenorrhea, a gynecological health problem that is frequently observed in adolescents and young adult women and often cannot be diagnosed is defined as pelvic pain associated with menstruation.

Providing analgesia without using pharmacological treatment is the leading aim of health care and can reduce drug-related complications. Therefore, nurses' awareness of the use of complementary and alternative medicine should be raised and the methods used should be based on evidence. Our search for studies in which the effects of listening to music and ice massage applied to the Hegu point on pain management in individuals with dysmenorrhea were investigated demonstrated that the number of such studies in the literature is not many. We think that the present study is important in terms of increasing the comfort levels of individuals with dysmenorrhea, basing the applications on evidence and contributing to the literature. It was conducted to compare the effects of ice massage applied to the Hegu point and music on pain and comfort levels in nursing students with dysmenorrhea.

DETAILED DESCRIPTION:
Dysmenorrhea, a gynecological health problem that is frequently observed in adolescents and young adult women and often cannot be diagnosed, is defined as pelvic pain associated with menstruation. The prevalence of dysmenorrhea is reported to vary between 50% and 90% in women of reproductive age. Dysmenorrhea and the symptoms accompanying dysmenorrhea cause significant economic losses by leading to both work and school absenteeism. Particularly in adolescents, due to dysmenorrhea, participation in sports and social activities is restricted, indicators of academic performance such as school absenteeism, school success, concentration, productivity are negatively affected, and thus their levels of general comfort and quality of life decrease. On the other hand, pharmacological treatment options used in the treatment of dysmenorrhea are very few. On top of this, the effectiveness of these treatment options is still debated. Since the medication used in the pharmacological treatment of dysmenorrhea has various side effects, using non-pharmacological treatments in addition to pharmacological treatment in the management of dysmenorrhea would be beneficial.

Cold application is one of the effective, simple, inexpensive and reliable non-pharmacological methods used to reduce pain, with few complications or no side effects. The Hegu point, the most important pain relief point of the body, can be stimulated in all painful conditions. Another low-risk and low-cost nonpharmacological method for standard care used in pain management is the music medicine.

This randomized clinical trial was designed to determine the effects of ice massage applied to the Hegu point and music on dysmenorrhea, compared to a control group that no intervention in women of 18 years or older from the the Faculty of Health Sciences at the Manisa Celal Bayar University, Manisa, Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Having menstruation regularly (between 21 and 35 days),
* Not using traditional and complementary treatments such as analgesics or massage during the application,
* Not having a diagnosed psychiatric problem and a history of endometriosis in the past,
* Not having infection and ovarian cyst / tumor, not having a neuropathic problem that might cause diabetes or nerve damage,
* Being over 18 years of age and agreeing to participate in the study.

Exclusion Criteria:

* Having hearing problems,
* Having connective tissue diseases,
* Having bleeding and coagulation disorders,
* Having fractures in the hand and arm to undergo therapy,
* Having sensitivity to cold,
* Using oral contraceptives.

Ages: 18 Years to 33 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — over 18 years
Enrollment: 129 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Questions about the menstrual characteristics of the students were asked using the Dysmenorrhea identification form | It took approximately 5-10 minutes to fill out the form.
  Questions about the menstrual characteristics of the students were asked using the Dysmenorrhea identification form developed by the researchers in line with the literature.
The intensity of pain experienced during the last menstrual period was asked using the Visual Analogue Scale (VAS | It took approximately 5-10 minutes to fill out the form.
  The intensity of pain experienced during the last menstrual period was asked using the Visual Analogue Scale (VAS). The highest pain score that can be obtained on the Visual Analogue Scale is 10 and the lowest is 0. The higher the score, the higher the pain intensity.
To evaluate dysmenorrhea severity using Functional and Emotional Dysmenorrhea Scale. | It took approximately 5 minutes to fill out the form.
  We asked them to determine the emotions they experienced on the first day of menstruation in accordance with the Functional and Emotional Dysmenorrhea Scale developed by Li et al. The minimum and maximum possible scores to be obtained from the scale are 14 and 70 respectively. The higher the score obtained from the Functional and Emotional Dysmenorrhea Scale is, the higher the functional and emotional disturbance levels of the individual affected by dysmenorrhea are In the second stage of the study, of the students, those who obtained ≥42 points from the Functional and Emotional Dysmenorrhea Scale and those who obtained ≥5 points from the Visual Analogue Scale were included in the study.
The Student Information Form | It took approximately 5 minutes to fill out the form.
  After the students who met the sample selection criteria and agreed to participate in the study were informed about the study, they were asked to fill in the Student Information Form.
  Questions about the sociodemographic and menstruation characteristics of the students were asked using the Student Information Form developed by the researchers in line with the literature.
Description of the students' comfort level. | It was evaluated on the first day of the menstrual cycle before the application. It took approximately 5-10 minutes to fill out the form.
  On the first day of the participating students' menstruation, prior to the application (when the pain started), General Comfort Questionnaire (GCQ) were filled in at the pre-test. The lowest and highest possible scores that can be obtained from the General Comfort Questionnaire are 1 and 4 respectively. While 1 point indicates that the level of comfort is low, 4 points indicate that the level of comfort is high.
To evaluate assessing menstrual pain characteristics. | It was evaluated on the first day of the menstrual cycle before the application. It took approximately 1-2 minutes to fill out the form.
  On the first day of the participating students' menstruation, prior to the application (when the pain started), Dysmenorrhea Follow-up Form were filled in at the pre-test. The questions in the form are as follows: time of onset of menstruation pain, the region where menstruation pain intensifies, the frequency of menstruation pain, the presence of complaints accompanying menstruation pain, the benefit of the method applied to relieve menstruation pain.
To evaluate the severity of pain secondary to dysmenorrhea with the Visual Analogue Scale (VAS) | up to 2 days
  We asked them to determine the severest pain score they felt on the first day of menstruation according to the Visual Analogue Scale (VAS).The highest pain score that can be obtained on the Visual Analogue Scale is 10 and the lowest is 0. The higher the score, the higher the pain intensity.
To evaluate the effect of Hegu point ice massage in reducing the pain severity secondary to dysmenorrhea through a Visual Analogue Scale (VAS). | up to 2 days
  The Hegu point of the participating students was detected with the acupuncture point finder.
  Ice cubes whose dimensions were 2x2x2 cm were wrapped with gauze and placed in a plastic bag. To prevent damage to the tissue and to ensure the sustainability of the movement, Vaseline® jelly was spread on the application area. We applied 2 minutes of ice massage 7 times at 15-second intervals. Melted ice cubes were replaced with new ones. As soon as the application was over, 30 and 60 minutes after the application, the participants' pain levels were assessed (Post-test). Pain intensity was measured with Visual Analogue Scale (VAS).The highest pain score that can be obtained on the Visual Analogue Scale is 10 and the lowest is 0. The higher the score, the higher the pain intensity. The procedure was performed once on the first day and once on the second day of menstruation.
To evaluate the effect of music medicine in reducing the pain severity secondary to dysmenorrhea through a Visual Analogue Scale (VAS). | up to 2 days
  Depending on their preference, each participant wearing personalized headphones was played instrumental music in the first and second day of menstruation for 30 minutes. As soon as the application was over, 30 and 60 minutes after the application, the participants' pain levels were assessed (Post-test). Pain intensity was measured with Visual Analogue Scale (VAS).The highest pain score that can be obtained on the Visual Analogue Scale is 10 and the lowest is 0. The higher the score, the higher the pain intensity. The procedure was performed once on the first day and once on the second day of menstruation.
To evaluate the effect of Hegu point ice massage in increasing comfort level. | It was evaluated on the second day of the menstrual cycle and after the application. It took approximately 5 minutes to fill out the form.
  On the second day of menstruation, the participants were asked to fill in the General Comfort Questionnaire (GCQ). The lowest and highest possible scores that can be obtained from the General Comfort Questionnaire are 1 and 4 respectively. While 1 point indicates that the level of comfort is low, 4 points indicate that the level of comfort is high.
To evaluate the effect of music medicine in increasing comfort level. | It was evaluated on the second day of the menstrual cycle and after the application. It took approximately 5 minutes to fill out the form.
  On the second day of menstruation, the participants were asked to fill in the General Comfort Questionnaire (GCQ). The lowest and highest possible scores that can be obtained from the General Comfort Questionnaire are 1 and 4 respectively. While 1 point indicates that the level of comfort is low, 4 points indicate that the level of comfort is high.
To determine the level of students being affected by dysmenorrhea. | It was evaluated on the second day of the menstrual cycle and after the application. It took approximately 5-10 minutes to fill out the form.
  On the second day of menstruation, the participants were asked to fill in the Effects of Dysmenorrhea Scale (EDS). It consists of 39 items and 11 sub-dimensions. Responses given to the items are rated on a 5-point Likert-type scale ranging from 1 to 5. The minimum and maximum possible scores to be obtained from the scale are 39 and 195 respectively. The higher the score obtained from the Effects of Dysmenorrhea Scale is, the higher the level of being affected by dysmenorrhea is.

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi PAKİŞ ÇETİN, Res Asis Dr, Principal Investigator — Celal Bayar University
Locations (1):
- Celal Bayar University, Manisa, Uncubozköy, Turkey (Türkiye)